CLINICAL TRIAL: NCT02535676
Title: Treatment of Negative Symptoms of Schizophrenia With Transcranial Direct Current Stimulation (tDCS): A Randomized, Double-blinded, Sham-controlled, Clinical Trial
Brief Title: Schizophrenia TreAtment With electRic Transcranial Stimulation
Acronym: STARTS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Instituto Bairral de Psiquiatria (Other); Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Leandro Valiengo, Medical Assistance, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 31063714.1.1001.0068
Record Dates: First submitted 2015-08-26; First posted 2015-08-28 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Schizophrenia
Keywords: schizophrenia; transcranial stimulation
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active tDCS (Active Comparator): Sham Comparator: Sham Stimulation In active stimulation, the anode is placed over the left dorsolateral prefrontal cortex and the cathode is placed over the temporo-parietal cortex with the Transcranial Direct Current Stimulation. The device will deliver a charge of 2mA for 20 minutes.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham tDCS (Sham Comparator): Sham Comparator: Sham Stimulation In active stimulation, the anode is placed over the left dorsolateral prefrontal cortex and the cathode is placed over the temporo-parietal cortex with the Transcranial Direct Current Stimulation. The device will deliver a charge of 2mA for 1 minute, after that the device will be automatically turned off for 19 minutes.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — The device will produce a direct current of 2 mA from one electrode to the other. In active stimulation, the device will be turned on for 20 min and in sham stimulation the device will be turned in 2 mA for one minute and will be automatically turned off the remaining 19 minutes. The sham or active mode is chosen by a numeric code.
  Other Names: Transcranial eletric stimulation

SUMMARY:
The aim of this study is to evaluate the therapeutic efficacy of tDCS (transcranial direct current stimulation) for treatment of negative symptoms in patients with schizophrenia. The proposed design is a clinical trial, randomized, double-blind, placebo-controlled study. Participants will receive ten sessions of active or sham stimulation in five consecutive days. 100 patients will be randomized into two groups (active tDCS vs sham tDCS) and will be assessed after the intervention: 2, 4, 6 and 12 weeks after. As objectives, the investigators expect to see a clinical improvement of negative symptoms through scales PANSS (Positive and Negative Syndrome Scale), Calgary, Auditory verbal hallucinations, SANS (Skills for Assessment of Negative Symptoms), and expect improvement on computerized cognitive tests. Another goal is to see improvement in biological markers related to schizophrenia, plasma and DNA will be stored.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia according to DSM-IV criteria and confirmed by the SCID
* Minimum score of 20 points in the sum of negative PANSS
* Stable antipsychotic medications

Exclusion Criteria:

* Unstable medical illness
* Uncontrolled pretreatment with rTMS or tDCS
* At least six months without being in ECT
* Benzodiazepines in doses of 10mg of diazepam
* Electronic or metal implants in the cephalic segment.
* Other mental disorders and dependence of substances

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-11; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change in subscale of PANSS | Repeated measures: 0, 2, 4 and 6 weeks (endpoint)
  Reduction of PANSS negative subscale (continuous measure) at 6 weeks

SECONDARY OUTCOMES:
Change in SANS | Repeated measures: 0, 2, 4, 6 and 12 weeks
  Reduction of SANS (continuous measure)
Change in Negative subscale of PANSS | 12 weeks
  Reduction of PANSS negative subscale (continuous measure)
Change in Auditory Verbal Hallucination Scale | Repeated measures: 0, 2, 4, 6 and 12 weeks
  Continuous measure

CONTACTS AND LOCATIONS:
Overall Officials: Leandro Valiengo, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Bulubas L, Goerigk S, Gomes JS, Brem AK, Carvalho JB, Pinto BS, Elkis H, Gattaz WF, Padberg F, Brunoni AR, Valiengo L. Cognitive outcomes after tDCS in schizophrenia patients with prominent negative symptoms: Results from the placebo-controlled STARTS trial. Schizophr Res. 2021 Sep;235:44-51. doi: 10.1016/j.schres.2021.07.008. Epub 2021 Jul 22. PMID 34304146
- [Derived] Valiengo LDCL, Goerigk S, Gordon PC, Padberg F, Serpa MH, Koebe S, Santos LAD, Lovera RAM, Carvalho JB, van de Bilt M, Lacerda ALT, Elkis H, Gattaz WF, Brunoni AR. Efficacy and Safety of Transcranial Direct Current Stimulation for Treating Negative Symptoms in Schizophrenia: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Feb 1;77(2):121-129. doi: 10.1001/jamapsychiatry.2019.3199. PMID 31617873
- [Derived] Valiengo L, Gordon PC, de Carvalho JB, Rios RM, Koebe S, Serpa MH, van de Bilt M, Lacerda A, Elkis H, Gattaz WF, Brunoni AR. Schizophrenia TreAtment with electRic Transcranial Stimulation (STARTS): design, rationale and objectives of a randomized, double-blinded, sham-controlled trial. Trends Psychiatry Psychother. 2019 Jun 19;41(2):104-111. doi: 10.1590/2237-6089-2018-0047. PMID 31241683